CLINICAL TRIAL: NCT05762653
Title: Morphological Features of the Pancreas in Patients With Type 2 Diabetes Mellitus: Correlation With Clinical Features of the Disease.
Brief Title: Morphological Pancreatic Features in Diabetes Mellitus Type 2
Acronym: PANDIAM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Clinico Universitario de Santiago (Other)
Responsible Party: Principal Investigator, J. Enrique Domínguez-Muñoz, Director of the Department of Gastroenterology, Hospital Clinico Universitario de Santiago
Other Study IDs: PAN-DM-01/2021
Record Dates: First submitted 2022-07-05; First posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: pancreatic fibrosis; endoscopic ultrasound; elastography; fecal elastase
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Endosonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: Cases are adult patients with type-2 diabetes, who undergo endoscopic ultrasound examination for any non-pancreatic indication.
  Interventions: Diagnostic Test: Endoscopic ultrasound
- Control: Controls are adult, non-diabetic patients, who undergo endoscopic ultrasound examination for any non-pancreatic indication.
  Interventions: Diagnostic Test: Endoscopic ultrasound

INTERVENTIONS:
Diagnostic Test: Endoscopic ultrasound — Evaluation of pancreatic fibrosis by endoscopic ultrasound and elastography. Evaluation of exocrine pancreatic function by fecal elastase-test and nutritional evaluation.
  Other Names: Fecal elastase test; Nutritional evaluation

SUMMARY:
Hypothesis: Type 2 diabetes mellitus is associated with pancreatic fibrosis that can be evaluated by minimally invasive imaging techniques. That fibrosis is associated with alteration of exocrine pancreatic function, defined as a reduced secretion of pancreatic enzymes and the development of nutritional deficiencies.

To test that hypothesis, a prospective, observational, cross-sectional, comparative, case-control study has been designed.

Pancreatic fibrosis will be evaluated by endoscopic ultrasound and quantitative elastography in cases (type-2 diabetes) and age-gender-matched controls without diabetes.

Pancreatic function will be explored by fecal elastase test and nutritional evaluation.

Calculated sample size is 94 patients (47 cases and 47 controls). Study period is 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years.
* Undergoing an upper endoscopic ultrasound for any indication other than pancreatic disease.
* Signed informed consent-
* Patients: Previous diagnosis of type-2 diabetes mellitus.
* Controls: Nondiabetic subjects, matched by age, gender, alcohol consumption, and smoking with patients.

Exclusion Criteria:

* History of pancreatic disease or surgery.
* History of upper gastrointestinal surgery.
* Diabetes type other than type-2.
* Severe cardiovascular or respiratory disease.
* Lack of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult diabetic (patients) and nondiabetic (controls) undergoing endoscopic ultrasound for indications other than evaluation of the pancreas due to suspected or known pancreatic disease.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Estimated)
Dates: Start 2022-02-03 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Degree of pancreatic fibrosis | Day 1
  Evaluation of the degree of pancreatic fibrosis by endoscopic ultrasound and elastography.
Degree of impairment of exocrine pancreatic function | Up to 7 days
  Quantification of fecal elastase and evaluation of the nutritional status

SECONDARY OUTCOMES:
Prevalence of pancreatic atrophy | Day 1
  Size of the pancreas as evaluated by endoscopic ultrasound
Factors associated with pancreatic fibrosis | Day 1
  Demographics and clinical data significantly associated with pancreatic fibrosis

CONTACTS AND LOCATIONS:
Overall Officials: J. Enrique Dominguez-Munoz, MD, PhD, Principal Investigator — University Hospital of Santiago de Compostela, Spain
Locations (1):
- Hospital Clinico Universitario de Santiago, Santiago de Compostela, A Coruña, Spain